CLINICAL TRIAL: NCT01136694
Title: Economic Burden in Adult Patients Diagnosed With Rheumatoid Arthritis (RA) Receiving Treatment With Biologic Disease-modifying Antirheumatic Drugs (bDMARDs)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-230
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients who are new bDMARD users
- RA patients who are existing DMARD users

SUMMARY:
The purpose of this study is to explore the differences in productivity loss and costs between patients being treated for rheumatoid arthritis (RA) with biologic disease-modifying antirheumatic drugs (bDMARDs) compared to patients treated with conventional DMARDs.

DETAILED DESCRIPTION:
Time Perspective: Prospective with some retrospective analysis of claims data

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a bDMARD or DMARD during the identification period (01 February 2009 - 31 July 2009)
* 18 years of age or older at the index year
* At least 12 months of continuous enrollment in a large commercial US health plan affiliated with i3 Innovus, including the at least 6 months and up to 12 months prior the index date (i.e., the pre-index period) and at least 6 months following the index date (i.e., the post-index (follow-up) period)
* Diagnosis of RA (reported on baseline survey)

Exclusion Criteria:

* Diagnosis of psoriasis, plaque psoriasis, or psoriatic arthritis (ICD-9 code 696.0x, or 696.1x), ankylosing spondylitis (720.0x), Crohn's disease (555.x), non-Hodgkins lymphoma (200.xx, 202.0x-202.2x, 202.7x-202.8x), or ulcerative colitis (556.x) in any position at any time during the 18-month identification period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Non-Probability Sample
Enrollment: 695 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patient-reported productivity loss using the Work Limitations Questionnaire (WLQ) | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)

SECONDARY OUTCOMES:
Direct and Indirect costs associated with lost productivity (as measured by WLQ) | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)
Healthcare utilization and costs (total and RA-related) | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)
Functionality (as measured by HAQ-DI) | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)
RA severity (as measured by RAPID3) | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)
Patient reported quality of life | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)
Patient reported treatment satisfaction | At baseline (6-12 months after starting index bDMARD; variable for DMARD) and at 6 months (12-18 months after starting index bDMARD; variable for DMARD)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm